CLINICAL TRIAL: NCT02205541
Title: Early Treatment With the Monoclonal C5 Antibody Eculizumab in Pediatric Patients Affected by Shiga-toxin Related Hemolytic and Uremic Syndrome: A Phase III Prospective Randomized Controlled Therapeutic Trial Versus Placebo
Brief Title: Eculizumab in Shiga-toxin Related Hemolytic and Uremic Syndrome Pediatric Patients - ECULISHU
Acronym: ECULISHU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC31/13/7052; PHRC 13-0060 (Other Grant/Funding Number: French Ministry of Health, PHRC 2013); 2014-001169-28 (EudraCT Number)
Record Dates: First submitted 2014-07-28; First posted 2014-07-31 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Hemolytic Uremic Syndrome of Childhood
Keywords: Eculizumab; Shiga-toxin; hemolytic and uremic syndrome; pediatric
MeSH Terms: conditions — Hemolytic-Uremic Syndrome | interventions — eculizumab; Solutions; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eculizumab (Experimental): 300mg concentrate for solution for infusion. According to the patient body weight, there will be 3 to 5 injections administered in IV infusion at D0, D7, D14, D21 and D28.
  Eculizumab (ECZ) will be administrated intravenously as a 30-minute injection.
  Interventions: Drug: Eculizumab
- Placebo (Placebo Comparator): Infusion of a solution with 5% glucose. The administration scheme will be the same as the Eculizumab arm : there will be 3 to 5 injections at D0, D7, D14, D21 and D28.
  Placebo will be administrated intravenously as a 30-minute injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eculizumab — According to the patient body weight, there will be 3 to 5 injections at D0, D7, D14, D21 and D28. According to the length of initial hospital stay, patients may have the remaining injections in the day ward of the recruiting center. Dosage of ECZ will be based on previous trials using ECZ in pediatric aHUS patients.
  ECZ or placebo will be administrated intravenously as a 30-minute injection
  Other Names: Soloris®
  Arms: Eculizumab
Drug: Placebo — According to the patient body weight, there will be 3 to 5 injections at D0, D7, D14, D21 and D28.
  ECZ or placebo will be administrated intravenously as a 30-minute injection
  Other Names: Solution with 5% glucose
  Arms: Placebo

SUMMARY:
The investigators aim to perform the first controlled randomized prospective study using ECZ in pediatric STEC-HUS. This is of great interest as there is still no efficient specific therapy in that potentially devastating disease.

Furthermore, published data concerning the use of ECZ in STEC-HUS are controversial, reflecting statistical bias in retrospective or uncontrolled studies, thus emphasizing the need for prospective studies.

DETAILED DESCRIPTION:
Hemolytic and uremic syndrome (HUS), characterized by thrombocytopenia, hemolytic anemia and acute renal failure (ARF), mainly affects children younger than 5 years old. Shiga-toxin (Stx) related HUS (STEC-HUS) is due to Stx secreting bacteria (mainly enterohemorrhagic Escherichia Coli strains). Acute phase of STEC-HUS is severe with at least 50% of affected children requiring dialysis, 20% presenting neurological involvement and 5% cardiac involvement. Mortality rates can reach 5% in pediatric series and long-term renal sequels have been reported in at least 30% of surviving patients. Apart from supportive care, no specific treatment (such as plasma exchange) has proven its efficacy in this life-threatening disease.

Recently, activation of the complement alternative pathway (CAP) has been demonstrated in STEC-HUS patients and experimental studies have highlighted that Stx induce CAP activation on human endothelial cells and platelet-leucocytes complexes, in addition to its direct cell toxicity inducing apoptosis, both processes ending up in microvasculature thrombosis. CAP activation has been demonstrated as the cause of atypical HUS (aHUS) and ECZ, a monoclonal C5 antibody, which inhibits the terminal complement complex (TCC) formation, can efficiently prevent evolution to end stage renal disease in aHUS patients. In 2011, Lapeyraque et al. reported its possible efficacy in 3 severe STEC-HUS pediatric patients. Nevertheless, in STEC-HUS, ECZ has only been used in uncontrolled studies, mostly during the 2011 German outbreak, with conflicting results. Considering the lack of therapy to prevent life-threatening complications and renal sequels in STEC-HUS and the logically expected efficacy of ECZ, controlled studies are mandatory. In recruiting centers, STEC-HUS patients with ARF will be proposed to enroll the trial with the exception of patients with multiorgan. After parental consent, patients will be randomized to receive either ECZ or a dextrose-based placebo in a single blinded fashion. According to the patient body weight, there will be 3 to 5 injections at day (D) 0, D7, D14, D21 and D28. According to the length of initial hospital stay, patients may have the remaining injections in the day ward of the recruiting center. Dosage of ECZ will be based on previous trials using ECZ in pediatric aHUS patients. We designed a single blinded study because patients treated with placebo who will develop severe multiorgan involvement will be switched to the ECZ arm. ECZ or placebo will be administrated intravenously as a 30-minute injection. In patients receiving hemodialysis, ECZ injection will be performed after a dialysis session. Before first injection, patients will receive a tetravalent meningococcal vaccine and an oral antibiotic prophylaxis to be continued up to 14 days after last injection.

This is a single blinded, phase III, randomized, multi-center controlled versus placebo clinical trial of eculizumab in STEC-HUS patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient (1 month-18 years old)
* Affected by STEC-HUS defined by :
* Thrombocytopenia (<150 000/mm3)
* Mechanic hemolytic anemia (Hemoglobin < 10g/dL, haptoglobin <LLN, lactate dehydrogenase (LDH) >upper limit of normal (ULN) and/or bilirubin > ULN, presence of schizocytes)
* ARF defined by an estimated Schwartz 2009 creatinin clearance <75ml/min/1,73m²
* With prodromal diarrhea and/or presence of an enterohemorrhagic strain of Escherichia Coli and/or identification of the Stx 1 or 2 genes in the stool sample or rectal swab
* Written consent of the 2 parents
* Female patients of childbearing potential must be practicing an effective, reliable and medically acceptable contraceptive regimen during the entire duration of the study and 5 months after the end of the participation.

Exclusion Criteria:

* Neonatal HUS
* Malignancy
* Known HIV infection
* Pregnancy or lactation
* Identified drug exposure-related HUS
* Infection-related HUS
* Known systemic lupus erythematosus or antiphospholipid antibody positivity or syndrome
* Patient already enrolled in a drug trial
* Patient with ongoing meningococcal infection
* Patient affected by aHUS or family history of aHUS
* STEC-HUS patient with severe multiorgan involvement at diagnostic:

  * Neurological involvement (seizures, coma, focal deficit) with signs of microangiopathy on cerebral Magnetic Resonance Imaging.
  * Cardiac involvement (cardiac failure, ischemic myocarditis, conduction or rhythm troubles)
  * Digestive involvement (severe pancreatitis defined by lipasemia>500UI/L, severe hepatitis defined by transaminase >x10ULN and/or prothrombin time<60%, hemorrhagic colitis, bowel perforation, rectal prolapsus)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
the duration in days of extrarenal epuration | From the inclusion date and assessed up to 13 months
  Extrarenal epuration means peritoneal dialysis or hemodialysis, and is assessed at each visit.

SECONDARY OUTCOMES:
Number of adverse events as a measure of Safety and tolerance of treatment injections (ECZ or placebo) | At each injection (treatment visits 2, 3, 4, 5, 6 at respectively day 0, 7, 14, 21, 28) and at each follow-up visit (7, 8, 9 respectively at month 2, 7, 13)
Adverse reactions related to the treatment (ECZ or placebo) | At each injection (treatment visits 2, 3, 4, 5, 6 at respectively day 0, 7, 14, 21, 28) and at each follow-up visit (7, 8, 9 respectively at month 2, 7, 13)
Duration of Acute Renal Failure (ARF) | Inclusion Visit (1 at day -3 to -1 ), treatment period (visits 2, 3, 4, 5, 6 respectively at day 0, 7, 14, 21, 28), follow-up period (visits 7, 8, 9 respectively at month 2, 7, 13)
  Duration of ARF will be evaluated as follow : urine output measurement, creatinin clearance estimated with the Schwartz 2009 assay (based on creatinin plasma levels), ionogram, proteinuria.
Renal sequels | At 1, 6 and 12 months after last injection of ECZ (follow-up visits 7, 8, 9)
  Renal sequels will be evaluated as follow : blood pressure, creatinin clearance, ionogram, proteinuria and microalbuminuria.
Hematological abnormalities | Inclusion Visit (1 at day -3 to -1), treatment period (visits 2, 3, 4, 5, 6 respectively at day 0, 7, 14, 21, 28), follow-up period (visits 7, 8, 9 respectively at month 2, 7, 13)
  * Duration (in days) of the thrombocytopenia
  * Duration (in days) of the hemolytic anemia
Blood parameters of Complement Alternative Pathway (CAP) | Inclusion visit (1 at day -3 to -1), Treatment visits (3, 4, 5, 6 at day 7, 14, 21, 28), follow-up visit (7 at month 2)
  Blood parameters of CAP will be evaluated with plasmatic dosages of the complement components C3 and CD46.
Inhibition of the Terminal Complement Complex (TCC) | Inclusion visit (1 at day -3 to -1), Treatment visits (3, 4, 5, 6 at day 7, 14, 21, 28), follow-up visit (7 at month 2)
  Inhibition of the TCC will be evaluated trough the CH50 assay and plasmatic free ECZ levels.
Incidence of extrarenal manifestations | Inclusion Visit (1 at day -3 to -1), treatment period (visits 2, 3, 4, 5, 6 respectively at day 0, 7, 14, 21, 28)
  * Neurological involvement (seizures, coma, focal deficit)
  * Cardiac involvement (cardiac failure, ischemic myocarditis, conduction or rhythm troubles)
  * Digestive involvement (pancreatitis, hepatitis, hemorrhagic colitis, bowel perforation, rectal prolapsus)
Mortality | Inclusion Visit (1 at day -3 to -1), treatment period (visits 2, 3, 4, 5, 6 respectively at day 0, 7, 14, 21, 28), follow-up period (visits 7, 8, 9 respectively at month 2, 7, 13)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Garnier, MD, Principal Investigator — University Hospital, Toulouse; Karine Brochard, Principal Investigator — University Hospital, Toulouse
Locations (18):
- France (18):
  - University Hospital, Amiens
  - University Hospital, Angers
  - University Hospital, Besançon
  - Pellegrin Hospital, Bordeaux
  - Morvan Hospital, Brest
  - University Hospital, Grenoble
  - Jeanne de Flandre Hospital, Lille
  - Mother and Child Hospital, Limoges
  - Women, Mother and Child Hospital, Lyon
  - La Timone Hospital, Marseille
  - University Hospital, Montpellier
  - Mother and Child Hospital, Nantes
  - Robert Debré Hospital, Paris
  - Trousseau Hospital, Paris
  - Necker Hospital, Paris
  - Anne de Bretagne University Hospital, Rennes
  - Purpan Children Hospital, Toulouse
  - Clocheville Hospital, Tours

REFERENCES:
- [Derived] Imdad A, Nelson JR, Tanner-Smith EE, Huang D, Gomez-Duarte OG. Interventions for preventing diarrhoea-associated haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2025 Apr 25;4(4):CD012997. doi: 10.1002/14651858.CD012997.pub3. PMID 40277027
- [Derived] Garnier A, Brochard K, Kwon T, Sellier-Leclerc AL, Lahoche A, Launay EA, Nobili F, Caillez M, Taque S, Harambat J, Michel-Bourdat G, Guigonis V, Fila M, Cloarec S, Djamal-Dine D, de Parscaux L, Allard L, Salomon R, Ulinski T, Fremeaux-Bacchi V, Morin C, Olivier-Abbal P, Colineaux H, Auriol F, Arnaud C, Kieffer I, Brusq C. Efficacy and Safety of Eculizumab in Pediatric Patients Affected by Shiga Toxin-Related Hemolytic and Uremic Syndrome: A Randomized, Placebo-Controlled Trial. J Am Soc Nephrol. 2023 Sep 1;34(9):1561-1573. doi: 10.1681/ASN.0000000000000182. Epub 2023 Jun 12. PMID 37303085
- [Derived] Groussolles M, Winer N, Sentilhes L, Biquart F, Massoud M, Vivanti AJ, Bouchghoul H, Rozenberg P, Olivier P, Desbriere R, Chauleur C, Perrotin F, Coatleven F, Fuchs F, Bretelle F, Tsatsaris V, Salomon LJ, Sananes N, Kayem G, Houflin-Debarge V, Schmitz T, Benoist G, Arnaud C, Ehlinger V, Vayssiere C; Groupe de Recherche en Gynecologie Obstetrique. Arabin pessary to prevent adverse perinatal outcomes in twin pregnancies with a short cervix: a multicenter randomized controlled trial (PESSARONE). Am J Obstet Gynecol. 2022 Aug;227(2):271.e1-271.e13. doi: 10.1016/j.ajog.2022.01.038. Epub 2022 Feb 3. PMID 35123930
- [Derived] Imdad A, Mackoff SP, Urciuoli DM, Syed T, Tanner-Smith EE, Huang D, Gomez-Duarte OG. Interventions for preventing diarrhoea-associated haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Jul 5;7(7):CD012997. doi: 10.1002/14651858.CD012997.pub2. PMID 34219224
- [Derived] Matrat L, Bacchetta J, Ranchin B, Tanne C, Sellier-Leclerc AL. Pediatric atypical hemolytic-uremic syndrome due to auto-antibodies against factor H: is there an interest to combine eculizumab and mycophenolate mofetil? Pediatr Nephrol. 2021 Jun;36(6):1647-1650. doi: 10.1007/s00467-021-05025-8. Epub 2021 Mar 28. PMID 33774745
- [Derived] Muff-Luett M, Sanderson KR, Engen RM, Zahr RS, Wenderfer SE, Tran CL, Sharma S, Cai Y, Ingraham S, Winnicki E, Weaver DJ, Hunley TE, Kiessling SG, Seamon M, Woroniecki R, Miyashita Y, Xiao N, Omoloja AA, Kizilbash SJ, Mansuri A, Kallash M, Yu Y, Sherman AK, Srivastava T, Nester CM. Eculizumab exposure in children and young adults: indications, practice patterns, and outcomes-a Pediatric Nephrology Research Consortium study. Pediatr Nephrol. 2021 Aug;36(8):2349-2360. doi: 10.1007/s00467-021-04965-5. Epub 2021 Mar 10. PMID 33693990